CLINICAL TRIAL: NCT06805448
Title: Intraglandular Treatment With Adipose-derived Mesenchymal Stem Cells in Patients With Xerostomia Due to Sjögrens Disease
Brief Title: Intraglandular Treatment With Adipose-derived Mesenchymal Stem Cells in Patients With Xerostomia Due to Sjögren's Disease
Acronym: ASSIX
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Joachim Hansen, Primary Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EU CT: 2024-516715-25-00; 2024-516715-25-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-21; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Sjorgren's Syndrome
Keywords: Mesenchymal stem/stromal cell; MSC; Advanced Therapy Medicinal Product (ATMP),; xerostomia; dry mouth; Sjogren's disease; Sjogren's syndrome; randomized clinical trial (RCT)
MeSH Terms: conditions — Xerostomia; Sjogren's Syndrome | interventions — Saline Waters

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Isotone sterile saline water
  Interventions: Drug: Saline Water (Control)
- MSC (Experimental): Allogeneic adipose-derived stem / stromal cells in 10% DMSO
  Interventions: Drug: MSC

INTERVENTIONS:
Drug: MSC — Allogeneic adipose-derived mesenchymal stromal / stem cells in 10% DMSO
  Arms: MSC
Drug: Saline Water (Control) — Isotonic sterile saline water
  Arms: Placebo

SUMMARY:
Living with dry mouth significantly impacts daily life, causing constant discomfort. It makes it harder to talk, eat solid food (increasing the risk of malnutrition), swallow, and sleep well. It also raises the risk of tooth decay. One common cause of dry mouth is Sjögren's Syndrome.

Sjögren's Syndrome is a common chronic autoimmune disease. In this disease, the immune system attacks the body's own saliva glands, reducing saliva production and leading to severe dry mouth and its associated symptoms.

Current treatments for dry mouth are temporary and only last a short time (from a few minutes to a few hours). Therefore, new treatment options are needed.

Research has shown that mesenchymal stem cells can be used to treat dry mouth with promising results. These stem cells can be injected into a vein or directly into the saliva glands. Although the exact mechanism is not fully understood, studies suggest that stem cells can positively affect the immune system, reduce inflammation, regenerate tissue, and reverse scarring.

This research group has been studying stem cell treatment for dry mouth for over 10 years and is internationally recognized. The group have conducted three studies where we injected stem cells into the saliva glands of patients with dry mouth due to radiation therapy for head or neck cancer. Results showed a 30%-50% increase in saliva production and a significant reduction in dry mouth symptoms. No studies have yet investigated injecting stem cells into the saliva glands of patients with dry mouth due to Sjögren's Syndrome. One study did inject stem cells into tear glands with promising results. Therefore, this study aim to investigate injecting stem cells into the saliva glands of patients with dry mouth due to Sjögren's Syndrome.

For this study, mesenchymal stem cells harvested from the fat tissue of healthy adult donors is used. This type of stem cell is better at reversing scarring and forming new blood vessels. The procedure is quick and has few side effects, and donors benefit from the fat removal. The fat is typically taken from the abdominal area. Donors are tested for various diseases to ensure they are healthy. Previous studies have shown that the treatment is safe with only a few temporary side effects.

The hypothesis is that injecting stem cells into the saliva glands of patients with dry mouth due to Sjögren's Syndrome will improve saliva production and reduce dry mouth symptoms. The study aims to determine if this treatment increases saliva production and reduces symptoms caused by dry mouth.

To test these hypotheses, the study will include:

1. The treatment itself with either stem cells or a placebo (sterile saline).
2. Multiple saliva tests to measure saliva production.
3. Saliva samples stored for later analysis to see if the saliva's ability to protect teeth and aid digestion changes after stem cell treatment.
4. A blood test to examine the immune system's response to the stem cell treatment.
5. A clinical examination to see if the stem cell treatment affects Sjögren's Syndrome symptoms elsewhere in the body.
6. Questionnaires to assess participants' perceptions of changes in dry mouth symptoms after treatment.

The treatment involves injecting either stem cells or a placebo into the two saliva glands near the jaw, guided by an ultrasound scan. The procedure takes 10 minutes.

Although stem cell treatment has been shown to be safe, safety will be monitored in this study. At all three visits, participants will be asked about any side effects, which will be categorized as serious or mild, and as treatment-related or not. Follow-up and treatment plans will be made for any side effects. Participants will also always have direct access to the treating doctor.

The study will be monitored by the Danish Medicines Agency and the GCP unit, which ensures that all rules and laws are followed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with SS according to the American College of Rheumatology/European League Against Rheumatism (ACR-EULAR) classification criteria for primary SjD (2)
2. Age equal or above 18 years
3. Persistent xerostomia for at least 3 months
4. Unstimulated whole saliva flow rate (UWS) of minimum 0.05 ml/min and maximum 3.0 ml/min
5. Capable and willing to receive proper information and to give written informed consent.

Exclusion Criteria:

1. Current intake of xerogenic medications such as anticholinergics, tricyclic antidepressants, opioids, and certain antihypertensive agents (23)
2. Presence of any other diseases of the salivary glands, e.g. xerostomia due to radiation
3. Previous submandibular gland surgery
4. Previous treatment with any type of stem cells in the salivary glands
5. Pregnancy or planned pregnancy within the 12 months study period
6. Breastfeeding
7. Tobacco smoking within the previous 6 months from screening visit
8. Have a current alcohol abuse (consumption must not exceed 10 units per week (Danish National board health alcohol guidelines (24))
9. Any other disease/condition judged by the investigator to be grounds for exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in unstimulated whole saliva flow rate by sialometry | From baseline to 4 months after treatment

SECONDARY OUTCOMES:
Change in stimulated whole saliva flow rate by sialometri | From baseline to 4 and 12 months after treatment
• Safety evaluated by number of serious adverse events (SAE), adverse advents (AE), and deaths | From baseline to 4 and 12 months after treatment
Quality of the whole saliva measured as changes in percentages in the concentration of electrolytes, total protein, alpha-amylase, and salivary IgA with Elisa assays | From baseline to 4 and 12 months after treatment
  The concentrations of the specific electrolyte, total protein and IgA will be compared to reference values.
Immune response measured by the development of donor specific antibodies | From baseline to 4 and 12 months after treatment
  Serum will be frozen until the end of the trial and all samples will be analyzed together. The blood samples will be analyzed for HLA class I and class II antibodies with the Luminex platform (Luminex 200 system or LABScan3D) and will be reported as HLA antibodies present/not present in the samples.
Lacrimal secretion measured by the Schirmers Test | From baseline to 4 and 12 months after treatment
• Changes in the gland morphology as assessed by ultrasound | From baseline to 4 and 12 months after treatment
  Measured as changes in the OMERACT US system
• Changes in ESSDAI | From baseline to 4 and 12 months after treatment
• Changes in ESSPRI | From baseline to 4 and 12 months after treatment
PROM: Xerostomia Questionnaire | From baseline to 4 and 12 months after treatment
  This PROM will be compared by converting to summary-scores ranging from 0-100.
PROM:Clinical Oral Dryness score. | From baseline to 4 and 12 months after treatment
  This outcome will be compared by converting to summary-scores ranging from 0-100
PROM: Summated Xerostomia Inventory. | From baseline to 4 and 12 months after treatment
  This outcome will be compared by converting to summary-scores ranging from 0-100

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Access to participant level-data and statistical code can be granted through a reasonable request to the corresponding author and subsequent approval from the relevant authorities.
Supporting Information: Study Protocol, SAP
Time Frame: Full protocol in available through CTIS (https://euclinicaltrials.eu/).
  IPD will be available after last patient's last visit
Access Criteria: Access to participant level-data and statistical code can be granted through a reasonable request to the corresponding author and subsequent approval from the relevant authorities.

REFERENCES:
- Available data/document: Study Protocol: 2024-516715-25-00 — https://euclinicaltrials.eu/